CLINICAL TRIAL: NCT02235207
Title: Effectiveness of Fustra-Exercise Program on Pain, Physical Fitness and Quality of Life in Female and Male Office Workers Suffering From Recurrent Neck and Low Back Pain - a Randomized Controlled Trial
Brief Title: Effectiveness of Fustra-Exercise Program in Neck and Low Back Pain
Acronym: FUSTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Fustra International Oy (Unknown)
Responsible Party: Principal Investigator, Jaana Suni, Research and develompment manager, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R14030
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Neck Pain; Low Back Pain, Recurrent
Keywords: sedentary work; musculoskeletal pain; neuromuscular exercise; physical fitness; quality of life; work ability
MeSH Terms: conditions — Neck Pain; Low Back Pain; Musculoskeletal Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular exercise (Experimental): The exercise group will participate in Fustra20 Neck & Back neuromuscular exercise program.
  Interventions: Behavioral: Neuromuscular exercise
- Control group (No Intervention): Participants are encouraged to continue there usual physical activity and exercise

INTERVENTIONS:
Behavioral: Neuromuscular exercise — Fustra20 Neck & Back is individually guided, graded neuromuscular exercise program which is conducted twice a week for 20 times. Each session lasts one hour. After 20 sessions participants are encouraged to continue exercising at home with a help of an individual home exercise plan including diary of compliance.
  The main targets are to
  * improve movement control in different posture and movements of the neck and back
  * improve flexibility with active functional movements
  * improve pelvic, spine and shoulder-neck stability using co-contraction of several muscle groups, and thus enhancing gross movement of the whole kinetic chain
  * improve muscular endurance of shoulder neck area, trunk, pelvis and lower extremities
  Arms: Neuromuscular exercise

SUMMARY:
The purpose of the study is to investigate the effectiveness of Fustra® exercise program in relieving recurrent pain in the neck or/and back, and thus improve quality of life in female and male office workers. The hypothesis is that neuromuscular exercise will improve control of posture and movement, neck shoulder and trunk flexibility, trunk muscular endurance and leg strength, and thus decrease intensity of pain by 30% compared to non-exercise group. In addition, financial feasibility of the exercise program and effects of training on quality of life and perceived work ability are studied.

DETAILED DESCRIPTION:
Neck and low back pain (LBP) are the two major reasons for visiting a physician and they cause significant sickness absence from work. Neuromuscular exercise of at least moderate intensity is the only mode of therapeutic exercise, which has been shown to be effective in relieving pain and disability in recurrent or chronic neck and LBP.

This study examines the effects of a standardized exercise program Fustra20 Neck & Back applied individually by educated exercise leaders in about 30 private sports clubs located in different parts of Finland. The target is to have 5-6 participants in each club. Recruitment began with advertisements in two national level newspapers. Interested individuals were asked to contact UKK Institute (UKKI) by phone or e-mail. In addition, the website of UKKI and the sports clubs are used to reach people more locally. Structured telephone interview is conducted to screen the eligible participants. Two researchers select the participants according to eligibility criteria.

Accepted participants are invited to the study by personal e-mail including the detailed announcement of the study and approval papers to be signed in. The tester of each sport club, responsible for conducting the fitness measurements (baseline, 3 months, 12 months) will receive text message from UKKI including names and phone numbers of accepted study participants. After that UKKI sends similar type of text message to each Fustra exercise leaders including only those participants that were randomly allocated to exercise group.

The exercise group will participate in individually guided, graded exercise twice a week for 20 times. Each session lasts one hour. Fustra exercise leaders have a personal diary for each participant, where they make notes on compliance and contents of each exercise session. After 20 sessions participants are encouraged to continue exercising at home with a help of an individual home exercise plan including diary of compliance.

Participants allocated to control group are asked to continue their usual physical activity and exercise habits. After the final measurements at 12-month they have a possibility to participate to Fustra20 Neck & Back exercise for five times.

ELIGIBILITY:
Inclusion Criteria:

* age 30-50 years
* sedentary "office" worker sitting at least 6 hours per day
* rating of neck pain or low back pain in the past four weeks is at least 3 in 10 point scale (1-10)
* number of pain episodes (neck/back) in the past year is at least 2

Exclusion Criteria:

* chronic pain (neck/back) defined as continuous pain over 1 year
* serious former neck injury (fracture, surgery, whiplash, protruded disc)
* serious former back injury (fracture, surgery, protruded disc)
* engaged in neuromuscular exercise 3 times a week or more
* engaged in competitive sports
* pregnant

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in the intensity of pain in the neck or/and low back | Baseline, 12 months
  Visual analog scale (line 0-100) filled in electronically (Webrobol) for past 4 weeks assessed separately for neck and low back pain

SECONDARY OUTCOMES:
Change in the intensity of pain in the neck or/and low back | Baselilne, 3 months
  Visual analog scale (line 0-100) for past 4 weeks filled in electronically (Webrobol) assessed separately for neck and low back pain and
Change in musculoskeletal fitness index | Baselilne, 3 months
  Fitness index is computed based on age and sex specific norm-reference values of 5 standardized tests assessing balance, shoulder neck mobility, trunk flexibility, ability to stabilize trunk and lower extremity endurance strength.

OTHER OUTCOMES:
Change in the quality of life | Baseline, 12 months
  RAND 36 with six subscales
Changes in objectively measured physical activity and sedentary behaviour | Baseline, 12 months
  Accelerometer assessment for 7 days with simultaneous diary recordings on specific exercise
Changes in fear avoidance beliefs | Baseline, 12 months
  Fear Avoidance Questionnaire (FABQ) filled in electronically

CONTACTS AND LOCATIONS:
Overall Officials: Jaana H Suni, PhD, Principal Investigator — UKK Institute
Locations (1):
- UKK Institute for Health Promotion Research, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No